CLINICAL TRIAL: NCT07028957
Title: Effectiveness of Low Volume Versus High Volume of Local Anesthetic in Ultrasound Guided Combined Supraclavicular and Interscalene Block for Upper Limb Surgery; A Randomized Controlled Double Blinded Study.
Brief Title: Effectiveness of Low Volume Versus High Volume of Local Anesthetic in Ultrasound Guided Combined Supraclavicular and Interscalene Block for Upper Limb Surgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Misr University for Science and Technology (Other)
Responsible Party: Principal Investigator, Emad Lotfy Mohammed Ahmed, Lecturer of anesthesia & pain management, Misr University for Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2022/0085
Record Dates: First submitted 2025-06-11; First posted 2025-06-19 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Analgesia, Postoperative; Complications of Treatment
Keywords: Low volume local anesthetic for brachial plexus block; High volume local anesthetic; brachial plexus blocks; Ultrasound guided
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: randomized controlled double blinded study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (n=20); Low volume Local anesthetic (15-20 ml) (Experimental): 20 patients, will receive ultrasound guided combined Supraclavicular Block (SCB) with 7-10 ml (3.5-5 ml bupivacaine 0.5% plus 3.5-5 ml lidocaine 2%) and Interscalene Block (ISB) with 7-10 ml (3.5-5 ml bupivacaine 0.5% plus 3.5-5 ml lidocaine 2%).
  Interventions: Procedure: Group A; Low volume local anesthetic in Ultrasound guided combined Supraclavicular and Interscalene block for Upper limb surgery
- Group B: ( n=20); High volume local anesthetic ( 30-40ml) (Active Comparator): 20 patients, will receive ultrasound guided combined Supraclavicular Block (SCB) with 15-20 ml (7.5-10 ml bupivacaine 0.5% plus 7.5-10ml lidocaine 2%) and Interscalene Block (ISB) with 15-20 ml (7.5-10 ml bupivacaine 0.5% plus 7.5-10 ml lidocaine 2%).
  Interventions: Procedure: Group B; High volume local anesthetics (30-40ml) ultrasound guided combined Supraclavicular Block (SCB) and Interscalene Block (ISB)

INTERVENTIONS:
Procedure: Group A; Low volume local anesthetic in Ultrasound guided combined Supraclavicular and Interscalene block for Upper limb surgery — Group A; will receive ultrasound guided combined Supraclavicular Block (SCB) with 7-10 ml (3.5-5 ml bupivacaine 0.5% plus 3.5-5 ml lidocaine 2%) and Interscalene Block (ISB) with 7-10 ml (3.5-5 ml bupivacaine 0.5% plus 3.5-5 ml lidocaine 2%).
  Arms: Group A (n=20); Low volume Local anesthetic (15-20 ml)
Procedure: Group B; High volume local anesthetics (30-40ml) ultrasound guided combined Supraclavicular Block (SCB) and Interscalene Block (ISB) — Group B; High volume local anesthetics in ultrasound guided combined Supraclavicular Block (SCB) with 15-20 ml (7.5-10ml bupivacaine 0.5% plus 7.5-10 ml lidocaine 2%) and Interscalene Block (ISB) with 15-20 ml (7.5-10 ml bupivacaine 0.5% plus 7.5-10 ml lidocaine 2%).
  Arms: Group B: ( n=20); High volume local anesthetic ( 30-40ml)

SUMMARY:
The aim of this study is to evaluate the effectiveness of low versus high volumes of local anesthetic in ultrasound-guided combined supraclavicular block (SCB) and interscalene block (ISB) for upper limb surgery. This randomized, controlled trial will assess the analgesic effectiveness of low-volume local anesthetic in these blocks.

We hypothesize that a low volume will provide similar analgesic effects to a high volume, with fewer complications. The study will involve 40 adult ASA I and ASA II patients undergoing upper limb surgery, divided into two groups: Group A (low volume) and Group B (high volume).

The primary outcome will compare intraoperative and postoperative analgesic effects of different volumes.

The secondary outcome will evaluate complications related to local anesthetics (toxicity) and injection techniques (e.g., phrenic nerve palsy, pneumothorax, hematoma).

DETAILED DESCRIPTION:
I. Study setting and location:

The study will be conducted in Souad Kafafi Universty Hospital - Misr University for Science and Technology ( MUST).

II. Study population:

Study will be conducted on (40) adult ASA І & ASA ІІ patients who will undergo Upper limb surgery in Souad Kafafi Universty Hospital - MUST University. Patients will be divided into two equal groups; Group A; Low volume of local anesthetic and Group B; High volume of local anesthetic in Ultrasound guided combined supraclavicular and interscalene block.

III. Eligibility Criteria:

1. Inclusion criteria:

   The study will recruit 40 ASA physical status I, II patients of both sexes, 18 - 65 years old presented for Upper limb surgery.
2. Exclusion criteria:

1. Refusal of patients to participate. 2. History of allergic reactions to local anesthetics. 3. Bleeding disorders with INR > 1.5 and/or platelets < 50 000. 4. Rash or signs of infection at the injection site. 5. Emergency procedure. 6. ASA ІІІ to VI patients.

IV. Study Procedures

1. Randomization An online randomization program will be used to generate random list and to allocate patients into two study groups: Low volume Local anesthetic group A (n=20) and High volume Local anesthetic group B (n=20) in Ultrasound guided combined supraclavicular and interscalene block for Upper limb surgery . Random allocation numbers will be concealed in opaque closed envelops. The patient and investigator performing the block and assessing study outcomes will all be blinded to the study group allocation.
2. Study Protocol:

Following approval from research and ethical committee of Faculty of Medicine, MUST University, The study will recruit forty ASA physical status I, II patients of both sexes, 18 - 65 years old, who will undergo upper limb surgery. A written informed consent from patients will be provided preoperatively.

Exclusion criteria of this study will be; refusal of the patient, trauma survey on head neck, chest and abdomen should be free, patient with neurological deficits involving upper limb, bleeding tendency, anticoagulation therapy, patients with allergy to local anesthetics, local infection at the injection site, patients on sedative or antipsychotic drugs and body mass index (BMI) > 35.

Group A: 20 patients, will receive ultrasound guided combined Supraclavicular Block (SCB) with 7-10 ml and Interscalene Block (ISB) with 7-10 ml.

Group B: 20 patients, will receive ultrasound guided combined Supraclavicular Block (SCB) with 15-20 ml and Interscalene Block (ISB) with 15-20 ml.

The primary outcome of this study will be to compare the analgesic effects (intraoperative and postoperative) of different volumes of local anesthetic in Ultrasound guided combined SCB with ISB for upper limb surgery.

The secondary outcome will be to assess complications of local anesthetic and techniques of injection All patients will be subjected to systematic preoperative assessment including history, examination, and investigations. Visual analogue scale score (VAS) (0-10) will be explained to all candidates where zero corresponds to no pain and 10 is indicative of the worst unbearable pain.

Patient positioning and preparation for the block:

On arrival to the preparation room: A peripheral IV cannula (18 G) will be inserted in the contralateral upper limb (non-operable limb); premedication using 2 mg midazolam IV.

Patients will be transferred to the operating room where basic monitoring (Electrocardiography (ECG), Non- invasive Blood Pressure (NIBP) and pulse oximetry (SpO2) will be attached. Baseline heart rate, blood pressure, oxygen saturation and respiratory rate will be recorded as pre-block values.

The patient will be placed in supine position with the head turned 45 degrees to the contralateral side. For the ultrasound-guided supraclavicular block, an ultrasound machine (Mindray China DC-N2-Diagnostic Ultrasound System) and a 10-14 MHz linear type probe will be used. After skin preparation and local anesthetic infiltration of skin, the supraclavicular fossa will be scanned to locate the subclavian artery, first rib, pleura and brachial plexus, then a 22 gauge, 9 cm, echogenic needle (B. Braun) will be advanced from lateral to medial in plane with the probe. The needle will be advanced towards the upper trunk and the "corner pocket" where the lower trunk commonly lies and the local anesthetics will be injected.

For ultrasound-guided Interscalene block, the ultrasound transducer will be placed in the axial, oblique plane at the level of the cricoid cartilage to obtain the transverse view of the brachial plexus. Nerves in the Interscalene groove appear hypoechoic, distinctly round or oval, and will be located between the anterior and middle scalene muscles. 9 cm 22 G needle will be inserted at the outer end of the ultrasound transducer after local anesthetic infiltration of the skin. The needle will be advanced in plane with the transducer; then injection will be done toward C5, C6 and C7 cervical nerve roots.

After injection of local anesthetic the patients will be observed for the onset of both sensory and motor blockade and duration of analgesia (first request of analgesic) in both groups.

Postoperative assessment and analgesic regimen:

VAS score of pain will be assessed immediately postoperative in the PACU and every 6 hours for 24 hours.

The time to the first request of rescue postoperative analgesic will be "the time interval between the onset of block and the first request to postoperative analgesia". When patients first complain of pain "1st analgesia request".

In the postoperative period if patients start to complain (VAS >3); rescue analgesia will be given in the form of pethidine 0.5-1 mg/kg/6hours, paracetamol (Perfalgan®) 1gm IV drip/6 hours and ketorolac 30mg IV/8 hours, till VAS score become ≤ 3.

V. Study outcomes

1. Primary outcome Post-operative pain score by VAS scale.
2. Secondary outcome(s)

   * Time to first request of postoperative rescue analgesics.
   * Perioperative hemodynamic parameters.
   * Incidence of perioperative complications.

Sample size Sample sizing will be based on results obtained from previous studies. Calculation of the sample size revealed that at least 18 patients in each group were needed to detect a difference in pain score and to detect the importance of Analgesia in reduction of pain in compliance as small as 1.5 times its standard deviation (SD) with a power of 0.9 and a significance level of 0.05. The sample size was increased by two patients in each group (20 patients in each group) to compensate for misinterpretations of pain score in each group.

Statistical analysis The Statistical Package of Social Science software program (SPSS), version 21 (Chicago, IL, USA) will be used for all statistical comparisons. Continuous quantitative normally distributed data will be expressed as means and standard deviations (SD), while non-normally distributed data will be expressed as median and range. Qualitative nominal data will be expressed by percentage.

After testing for normality, continuous variables will be compared using t-test or Mann-Whitney U test as appropriate. Categorical variables will be compared using Chi- squared test or Fisher's exact test as appropriate. correction. A pvalue <0.05 will be considered statistically significant

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 65 of both sexes
* ASA classification I or II
* Scheduled for upper limp surgery
* Will be randomized 1:1 into two groups; group A; low volume local anesthetics (15-20ml) and group B; high volume local anesthetics (30-40 ml).

Exclusion Criteria:

* Patients who refuse participation.
* Have allergies to local anesthetics.
* Phrenic nerve dysfunction.
* Chronic opioid use.
* ASA III or higher classification.
* Coagulopathy (bleeding disorders with INR > 1.5 and/or platelets < 50 000)
* Severe chronic obstructive pulmonary disease.
* Local infection at the injection site

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-06-30 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Analgesia | From time of injection to end of first 24 hours
  The primary outcome of this study will be to compare the analgesic and anesthetic effect of different volumes of local anesthetic in Ultrasound guided combined SCB with ISB for upper limb surgery. measured by Visual analogue scale score score (VAS) (0-10; with 0 means no pain and 10 means most severe pain).

SECONDARY OUTCOMES:
complications of local anesthetic | From time of injection to end of surgery
  Signs of local anesthetics toxicity
complications of technique of injection | From time of injection to end of 24 hours postoperative
  Complications of the technique; pneumothorax, hematoma, phrenic nerve palsy...( yes/No)
Heart Rate (HR) beat/minute | before induction of anesthesia and every 15 minutes till end of surgery
  measuring the heart rate before anesthesia, after induction of analgesia and every 15 minutes during surgery to detect any changes in the patients HR in both groups
Mean Arterial Blood Pressure ( MAP)( mmHg) | Before anesthesia, after induction of analgesia and every 15 minutes during surgery
  measuring the mean arterial pressure (MAP) before anesthesia, after induction of analgesia and every 15 minutes during surgery to detect any changes in the patients MAP in both groups

CONTACTS AND LOCATIONS:
Overall Officials: Hossam S. El Din El Ashmawi, Prof. of anesthesia and pain, Study Chair — Cairo University
Locations (1):
- Souad Kafafi University Hospital (SKUH), faculty of medicine, Misr University for Science and Technology (MUST), Giza, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Demographic Information: Age, sex, race, and other relevant demographic details.
  Baseline Characteristics: Health status, medical history, and any pre-existing conditions prior to the trial.
  Treatment Assignment: Information on the intervention or treatment each participant received.
  Outcome Measures: Data on primary and secondary outcomes as defined in the trial protocol.
  Adverse Events: Reports of any side effects or adverse events experienced by participants during the trial.
  Follow-up Data: Information collected during follow-up periods, including long-term outcomes.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: from 01/02/2026 to 31/03/2026
Access Criteria: Researchers:
  Who: Academic researchers, industry scientists, and regulatory agencies. What: Full IPD, including demographic data, treatment assignments, and outcome measures.
  How: Through data sharing platforms or repositories after submitting a research proposal and obtaining necessary approvals.
  Regulatory Authorities:
  Who: Agencies like the FDA or EMA. What: Full IPD and supporting documentation for oversight and review. How: Direct access during the review process of clinical trial applications.
  Data Sharing Initiatives:
  Who: Collaborating institutions and consortia. What: Aggregated or anonymized IPD for meta-analyses or systematic reviews. How: Via established partnerships and shared databases.
  Public and Patient Advocacy Groups:
  Who: Organizations seeking to promote transparency. What: Summary data and aggregated results, but not individual-level data. How: Through publicly available reports or dashboards.

REFERENCES:
- [Background] Falyar CR, Grossman EC. Ultrasound-guided interscalene-supraclavicular block for an intramedullary nailing of a pathologic humeral fracture: practical application of ultrasound-guided regional anesthesia. AANA J. 2014 Jun;82(3):219-22. PMID 25109160
- [Background] Hadzic A. Hadzic's Textbook of Regional Anesthesia and Acute Pain Management. 2nd ed. New York: McGraw-Hill; 2017. p. 44.
- [Background] Fredrickson MJ, Krishnan S, Chen CY. Postoperative analgesia for shoulder surgery: a critical appraisal and review of current techniques. Anaesthesia. 2010 Jun;65(6):608-624. doi: 10.1111/j.1365-2044.2009.06231.x. PMID 20565394